CLINICAL TRIAL: NCT07045857
Title: Recurrence of H Pylori : Incidence and Influential Factors in Sohag Government.
Brief Title: Recurrence of H Pylori : Incidence and Influential Factors.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Tomas Wagih Thabet, Resident, Internal Medicine Department, Faculty of Medicine, Sohag University, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med--25-5-11MS
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- follow up of patients that had H. Pylori infection and recieved medical treatment for recurrence (Other): follow up of patients that had H. Pylori infection and recieved medical treatment for recurrence and influential factors for recurrence
  Interventions: Behavioral: follow up of patients that had H. Pylori infection and recieved medical treatment for recurrence

INTERVENTIONS:
Behavioral: follow up of patients that had H. Pylori infection and recieved medical treatment for recurrence — follow up of patients that had H. Pylori infection and recieved medical treatment for recurrence and influential factors for recurrence

SUMMARY:
This study aims to determine recurrence rates, identify influential factors, investigate key factors that contribute to recurrence, evaluate treatment effectiveness and to assess the efficacy of different eradication regimens and their role in reducing recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old.
* H. pylori infection: Confirmed by endoscopy, biopsy, or non-invasive tests (e.g., urea breath test, stool antigen test).
* Symptoms: Presence of dyspepsia, peptic ulcer disease, or other H. pylori-related symptoms.
* Laboratory tests: Normal liver and kidney function, and no significant abnormalities in blood counts.

Exclusion Criteria:

* Patients receiving eradication therapy in the past taking proton pump inhibitors,, H2 blockers ,,bismuth ,, antibiotics or other medications that interfere with the result of the examination in the recent 4 weeks.
* Gastrointestinal disorders: Severe gastrointestinal disorders (e.g., gastric cancer, inflammatory bowel disease ,gastric or duodenal ulcer with current or recent bleeding , or clinical significant gastrointestinal bleeding within 4 weeks of randomization).
* Malignancies: Active or recent malignancies.
* Severe comorbidities: Unstable or severe comorbidities (e.g., heart failure, liver cirrhosis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
recurrence of H. Pylori infection in patients who recieved medical treatment | 4 weeks after successful medical treatment
  H. Pylori antigen in stool

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Mitchell HM, Hu P, Chi Y, Chen MH, Li YY, Hazell SL. A low rate of reinfection following effective therapy against Helicobacter pylori in a developing nation (China). Gastroenterology. 1998 Feb;114(2):256-61. doi: 10.1016/s0016-5085(98)70475-5. PMID 9453484
- [Background] Chen TS, Tsay SH, Chang FY, Lee SD. Triple therapy for the eradication of Helicobacter pylori and reduction of duodenal ulcer relapse: comparison of 1 week and 2 week regimens and recrudescence rates over 12 months. J Gastroenterol Hepatol. 1995 May-Jun;10(3):300-5. doi: 10.1111/j.1440-1746.1995.tb01097.x. PMID 7548807
- [Background] Anand PS, Kamath KP, Anil S. Role of dental plaque, saliva and periodontal disease in Helicobacter pylori infection. World J Gastroenterol. 2014 May 21;20(19):5639-53. doi: 10.3748/wjg.v20.i19.5639. PMID 24914323